CLINICAL TRIAL: NCT07192640
Title: PERIOPERATIVE USE OF INTRAVENOUS TRANEXAMIC ACID FOR HIGH BMI PATIENTS GOING THROUGH BARIATRIC SURGERIES
Brief Title: Intravenous Tranexamic Acid
Acronym: TXA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sabah Nageeb, anesthesia consultant, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KACS, KSA; KASC, KSA (Other: KING SALMAN SPECIALIST HOSPITAL , KSA, HAIL)
Record Dates: First submitted 2025-09-12; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Obese Patients; Obese Patients With Bariatric Surgery; Bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Intervention Model Description: After induction of anaesthesia tranexamic acid will be administered at the start of surgery to reduce intraoperative bleeding. loading dose of 10 mg/kg for high BMI patients who are undergoing bariatric surgery
  Control group of high BMI bariatrics patients will not receive TXA but will be operated by the same surgery team and homeostasis steps.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tranexamic group (Active Comparator): After induction of anesthesia tranexamic acid will be administered at the start of surgery to reduce intraoperative bleeding. loading dose of 10 mg/kg
  Interventions: Drug: After induction of anaesthesia tranexamic acid will be administered at the start of surgery to reduce intraoperative bleeding. loading dose of 10 mg/kg for high BMI patients who are undergoing bariatr
- control group (No Intervention): After induction of anaesthesia tranexamic acid will not be administered

INTERVENTIONS:
Drug: After induction of anaesthesia tranexamic acid will be administered at the start of surgery to reduce intraoperative bleeding. loading dose of 10 mg/kg for high BMI patients who are undergoing bariatr — This intervention will be applied for High-risk patients, with obesity, BMI more than 45, Preexisting cardiovascular condition, Hypertension, diabetes, or coagulation disorders, thyroid dysfunction and pulmonary disorders.
  Arms: tranexamic group

SUMMARY:
Tranexamic acid is a promising option for minimizing blood loss in high-risk bariatric surgery patients, particularly in those with obesity, diabetes, and other comorbidities. When used appropriately, TXA can reduce the need for blood transfusions, maintain hemodynamic stability, and lower the incidence of complications related to blood loss.

DETAILED DESCRIPTION:
The impact of TXA in high-risk individuals undergoing bariatric surgery is of increasing interest, especially given the inherent risks of bleeding and complications associated with these procedures. Bariatric surgery, particularly procedures like Roux-en-Y gastric bypass (RYGB) and sleeve gastrectomy, carries a risk of significant blood loss, which may be exacerbated in patients who are morbid obese or have underlying comorbid conditions such as hypertension, diabetes, or coagulation disorders.

TXA can effectively reduce intraoperative and postoperative blood loss by stabilizing fibrin clots, which is critical in preventing the need for transfusions and reducing surgical complications. A few studies have explored the use of TXA in bariatric surgery because of the fear of associated increased incidence of embolic complications.

ELIGIBILITY:
Inclusion Criteria:

* High-risk patients, with obesity, BMI more than 45,
* Patients with Preexisting cardiovascular condition, Hypertension, diabetes, or coagulation disorders, thyroid dysfunction and pulmonary disorders.

Exclusion Criteria:

* patients with active thromboembolic disorders.
* Patients with preexisting renal dysfunction,

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood Loss | "Perioperative"
  Intraoperative and postoperative Blood Loss will be calculated in the suction and wet gauzes by blood and the need for blood transfusion will be recorded

SECONDARY OUTCOMES:
postoperative risk of thromboembolism, infections, delayed wound healing, or longer hospital stays | pre-intervention/surgery""Postoperative "up to 1 week"
  The patients will be followed up for one week for possible incidence of side effects

CONTACTS AND LOCATIONS:
Locations (1):
- King Salman Specialist Hospital, Hail, KSA, Hail, Saudi Arabia

REFERENCES:
- Available data/document: Study Protocol — https://doi.org/10.1590/acb370702 — https://doi.org/10.1590/acb370702